CLINICAL TRIAL: NCT05049811
Title: An Overall Solution for Full-course Oral Anti-tumor Drug Services Based on Mobile Medicine
Brief Title: Effects of Mobile Medicine on Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FJZLYX002
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Cancer Pain
Keywords: mini program; self management; cancer pain
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a mini program trial group (Experimental): Pharmacists conducted a standardized education session to teach the participants how to operate the mobile phone, use mini program, assess pain. The participants in the trial group were asked to complete initial and final pain assessment questionnaires and Medication compliance on the mobile phones provided to them. Participants were encouraged to use mini program as much as possible to record their pain status.
  Interventions: Behavioral: mini program
- a control group (Sham Comparator): The control group received conventional pharmaceutical care. Initial and final pain and Medication compliance data were collected. Before the patient was discharged from the hospital, the clinical pharmacist conducted detailed medication education (including medication methods, prevention and treatment of adverse reactions, and precautions) and asked the patient to attempt to maintain a paper version of the pain diary.
  Interventions: Behavioral: conventional pharmaceutical care

INTERVENTIONS:
Behavioral: mini program — To design, construct, and test the mini program in patients managing cancer pain
  Other Names: "yao nin you wo "
  Arms: a mini program trial group
Behavioral: conventional pharmaceutical care — Regular education includes medication guidance from doctors, nurses and pharmacists.
  Arms: a control group

SUMMARY:
With the existing medical system and insufficient medical resources in China, we developed a mini program. a pain management mini app can be useful and appreciated by patients and health care professionals, making it a good choice for the management of cancer pain in our country . our study want to develop and test the mini program for pain management among Chinese cancer patients in or discharged from hospital treatment.

DETAILED DESCRIPTION:
Healthcare interventions delivered via personal mobile device have been shown to be acceptable to users, who have identified benefits such as convenience, access to personalized information, greater awareness of own health. Integrating mini program into the cancer pain care may be an effective strategy to improve cancer pain patients self-management.

To design, construct, and test the mini program in patients managing cancer pain, evaluate the total remission rate of pain and the improvement in medicine compliance to improve pain management for cancer pain patients, and assess patient acceptance of the mini program.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older;
* Be able to read Chinese and use a mobile phone;
* Histologically or cytologically confirmed solid tumor;
* Diagnosed chronic cancer pain
* Could understand the study process and evaluation, agreed to participate in the trial, and signed the informed consent form.

Exclusion Criteria:

* Illiterate person;
* Incompetence;
* Inability to complete the pain assessment;
* Participation in any other therapies or other study protocols that may have an impact on pain intensity, which were the main outcomes of this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change in pain score | Change from baseline at four weeks after discharge
  Comparison of pain score of cancer pain patients with or without mini program. Pain score will be assessed by using numeric rating scale (NRS). An NRS allows a person to describe the intensity of his/her pain as a number usually ranging from 0 to 10, where "0" means "no pain" and "10" means pain as "bad as it could be."

SECONDARY OUTCOMES:
Change in medication adherence | Change from baseline at four weeks after discharge
  The investigators will measure the change in medication adherence via Morisky Scale. Morisky Scale contains 4 questions, and the total score ranges from 0 to 4 with lower scores indicating higher adherence.
Incidence of adverse events | Up to four weeks after discharge
  Adverse events will be assessed throughout the study according the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event (CTCAE) Version 4.0. Number of subjects who experienced an adverse event in this study is presented.
Change in quality of life | Change from baseline at four weeks after discharge
  Comparison of quality of life of cancer pain patients with or without mini program. Quality of life is assessed using EuroQol- 5 Dimension (EQ-5D).

IPD SHARING:
Plan to Share IPD: No